CLINICAL TRIAL: NCT00642252
Title: Development and Validation of a Multi-Mineral Fluoride Mouthrinse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana Nanotech, LLC (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Robert L. Karlinsey, Managing Member, Indiana Nanotech, LLC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Nanotech Phase II April 2008
Record Dates: First submitted 2008-03-17; First posted 2008-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Dental Caries
Keywords: remineraliation; pre-existing white-spot (non-cavitated) enamel lesions
MeSH Terms: conditions — Dental Caries | interventions — Fluorides

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): 226 ppm fluoride + 30 ppm calcium 'prototype/new' mouthrinse
  Interventions: Drug: Fluoride
- A (Active Comparator): ADA-accepted over-the-counter 226 ppm fluoride mouthrinse (i.e. ACT, 226 ppm fluoride mouthrinse distributed by Chattem, Inc.)
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Fluoride — Over-the-counter level of fluoride (226 ppm) in a fluoride mouthrinse; FDA considers fluoride in a rinse formulation as a 'drug'; dosage is 10 mL per treatment.
  Other Names: ACT fluoride mouthrinse
  Arms: A
Drug: Fluoride — Over-the-counter level of fluoride (226 ppm) plus calcium (30 ppm) in a fluoride mouthrinse; FDA considers fluoride in a rinse formulation as a 'drug'; dosage is 10 mL per treatment.
  Other Names: New mouthrinse
  Arms: B

SUMMARY:
The primary goals of this project are to determine the anticaries benefits of a prototype multi-mineral mouthrinse containing 225 ppm fluoride and 30 ppm of a Ca through the remineralization of enamel white-spots (non-cavitated lesions). The selection of patients with pre-existing white-spot lesions will permit an opportunity to evaluate the efficacy of the multi-mineral mouthrinse in reminerzalizing and/or inhibiting progression of enamel white-spot lesions.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, panelists will be required to meet the following criteria:

1. Subjects must be 13 - 65 years of age;
2. Subjects must read and sign the Informed Consent prior to initiation of study procedures. All subjects will receive a copy of the signed Informed Consent;
3. Subjects must have a reasonable functional dentition, without a large number of missing teeth, and teeth #'s 22-27 present;
4. Have normal salivary gland function (unstimulated whole salivary flow rate equal to or greater than 0.25 ml/min and paraffin stimulated whole salivary flow rate equal to or at least 1.0 ml/min);
5. Subjects must be willing to participate in the study, be able to follow the study directions, be willing to return for all specified visits at their appointed time, and to use the product as per instructions;
6. Subjects must be in good general health based on medical history and oral soft and hard tissue examination.

Exclusion Criteria:

Criteria that will not permit participation in this study will be as follows:

1. Any subject who is pregnant or lactating - based on oral interview only - as pregnancy may interfere with the outcome of the study;
2. Any subject who has a systemic health condition such as diabetes that could affect the outcome of the study at the discretion of the examiner;
3. Any subject who has an oral condition, such as excessive, untreated dental caries, periodontal disease, chronic dental neglect, or any oral pathology including xerostomia determined by oral examination and subject history that in the opinion of the dental examiner could affect the outcome of the study;
4. Any subject who has full dentures, or full orthodontic appliances. No use of nightguards will be permitted during the study period;
5. Any subject who uses oral care products (other than those permitted) during the treatment or wash-out periods;
6. Any subject with an immunological disorders such as HIV positive, AIDS, and systemic Lupus Erythematosis;
7. Any subject concurrently participating in another clinical study;
8. Any subject currently taking antibiotics or other medications, which in the opinion of the Investigator/Examiner might influence the study outcome;
9. Any subject with a history of sensitivity to oral products or allergies to ingredients in the products;
10. Any subject who fails to keep any of their scheduled appointments.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Remineralization of non-cavitated enamel lesions. | baseline, 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: George K Stookey, PhD, Study Director — Indiana Nanotech
Locations (1):
- Crispus Attucks Medical Magnet High School, Indianapolis, Indiana, United States